CLINICAL TRIAL: NCT04228861
Title: Investigation of Colonization of Streptococcus Mutans, Lactobacillus Spp. and Candida Spp. in Oral Microflora in Infancy and Transmission From the Parent to the Infant
Brief Title: Investigation of Oral Microflora of Infants
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Zehra Beyza Erel, research assistant, Inonu University
Other Study IDs: 963
Record Dates: First submitted 2020-01-07; First posted 2020-01-14 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Streptococcus Mutans
Keywords: Familial transmission; Candida; Lactobacillus; S. mutans; newborn
MeSH Terms: conditions — Torulopsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — salivary
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The placement of cariogenic microorganisms in oral microflora is an important factor in dental caries. The aim of this study is to research from whom, when and how the cariogenic microorganisms are first transmitted to the infant. The investigators investigated of colonization of Streptococcus mutans, Lactobacillus spp., and Candida spp. in oral cavities of infants and their transmission to the infants.

DETAILED DESCRIPTION:
Study sample size and design: When α = 0.05, 1-β (power) = 0.80 were taken to determine the sample volume, it was calculated that at least 46 babies should be sampled for 6 months to have an average amount of S. mutans change of 1.87 units. Considering the losses that may occur during the follow-up, the study was started by taking samples from 60 systemically healthy newborns.

The study commenced with 60 newborns and was completed with 47 infants due to losses during the follow-up. Oral swab samples were taken from 47 healthy infants within the first 24 hours after birth, at 1 month old and during the first tooth eruption. Saliva samples were taken from the mothers of all the infants and from the fathers of 20 of the infants in the last meeting.

Last interview with the parents, their oral examinations were performed, and their findings were processed as decayed (D), filled (F) and missing (M) teeth in accordance with the World Health Organization criteria, with the DMF (decayed, missing and filled) index being calculated. Furthermore, saliva samples were taken from the parents at the last interview. A questionnaire form including the sex of the infant, type of delivery, birth weight, and nutritional habits of the infant during the follow-up was filled in by gaining information from the parents on the first day and during the follow-ups.

Swab samples taken from infants with sterile swabs were transferred to the laboratory by placing sterile saline solution into dispensed 2 ml screw cap tubes. Sterile urine collection containers of 50 ml were used to collect saliva samples from the parents.

ELIGIBILITY:
Inclusion Criteria:

* none of the infants or their families had systemic disease

Exclusion Criteria:

* the infants or their families have systemic disease

Ages: 30 Minutes to 2 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study was conducted in two centers - Turgut Özal Medical Center and Malatya Training and Research Hospital. Between January and May 2018, healthy newborns born in these two hospitals were followed up.
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Acquisition of the oral streptococcus mutans in infants | first 24 hours after birth
  Counts of oral streptococcus mutans
Acquisition of the oral streptococcus mutans in infants | at 1 month old
  Counts of oral streptococcus mutans
Acquisition of the oral streptococcus mutans in infants | 4 to 12 months depending on the first tooth eruption.This period changed according to the growth rate of the baby
  Counts of oral streptococcus mutans

SECONDARY OUTCOMES:
Acquisition of the oral Lactobacillus and candida spp. in infants | first 24 hours after birth
  Counts of oral Lactobacillus and candida spp
Acquisition of the oral Lactobacillus and candida spp. in infants | at 1 month old
  Counts of oral Lactobacillus and candida spp
Acquisition of the oral Lactobacillus and candida spp. in infants | 4 to 12 months depending on the first tooth eruption.This period changed according to the growth rate of the baby
  Counts of oral Lactobacillus and candida spp

CONTACTS AND LOCATIONS:
Overall Officials: gülsüm duruk, Study Director — Inonu University; zehra b erel, Principal Investigator — Inonu University
Locations (1):
- Inonu university, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I can think of sharing after becoming a publication in a journal